CLINICAL TRIAL: NCT02263729
Title: Phase 1/2 Prospective Double-blind, Placebo-controlled Randomized Clinical Trial Using Losartan to Treat Grade II and III Hamstring Strains
Brief Title: Phase 1/2 Prospective Double-Blind Placebo-Controlled Randomized Clinical Trial of Losartan to Treat Grade II & III Hamstring Strains
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to difficulty identifying eligible participants and the expiration of funding.
Sponsor: James J. Irrgang (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); Wake Forest University (Other)
Responsible Party: Sponsor-Investigator, James J. Irrgang, PT, PhD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY19100320; W81XWH-14-2-0003 (Other Grant/Funding Number: US Army Medical Research Acquisition Activity)
Record Dates: First submitted 2014-09-26; First posted 2014-10-13 (Estimated); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Hamstring Injury
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Losartan (Active Comparator): Subjects will taken 50mg of losartan per day for 4 weeks
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): Subjects will be given placebo to replicate appearance of losartan pills. Placebo pill will be taken once per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — Cozaar
  Arms: Losartan
Drug: Placebo
  Arms: Placebo

SUMMARY:
The goal of this study is to determine safety and tolerability of Losartan when used for treatment of an acute grade II or III hamstring strain and determining the effect of losartan on recovery of hamstring muscle function. Subjects will be adults age 18 and older with grade 2 or 3 hamstring injury who participate in greater than 100 hours per year in Level 1 or Level 2 athletics or have a similar activities or physical work load (e.g. military personnel). Subjects will undergo examination, MRI, and functional assessment before, during, and after 4 weeks of losartan (50mg QD) or placebo.

ELIGIBILITY:
Inclusion Criteria

1. 18 years of age and older;
2. Have had grade II or III hamstring injury within the 7 days prior to enrollment;
3. Greater than 100 hours per year in Level I (football, basketball, or soccer) or Level II (racquet sports, skiing, manual labor occupations/heavy physical work) and activities that require running and sprinting;
4. Agree to take study medications as prescribed

Exclusion Criteria:

1. Have had previous hamstring injury on the same side or chronic symptoms;
2. Have an injury that requires surgical intervention (e.g. avulsion with associated bony involvement, grade III complete tears);
3. Have concurrent lower back symptoms;
4. Pregnant or breast feeding;
5. Is a smoker;
6. Has contraindications for Losartan therapy (hypersensitivity to Losartan, hepatic involvement);
7. Currently use angiotensin I converting enzyme inhibitor (ACEI)/ Angiotensin II receptor blocker (ARB);
8. Have hypertension (blood pressure greater than or equal to 140 mmHg systolic pressure or greater than or equal to 90 mmHg diastolic pressure);
9. Have hypotension (blood pressure less than or equal to 90 mmHg systolic pressure or less than or equal to 60 mmHg diastolic pressure);
10. Have orthostatic hypotension defined as a drop in systolic pressure greater than or equal to 2 0mmHg or a drop in diastolic blood pressure greater than or equal to 10 mmHg or reports of lightheadedness or dizziness upon standing;
11. Have diabetes mellitus, cardiovascular, renal or hepatic co-morbidities;
12. Sickle cell anemia/trait;
13. Have contraindications for MRI - including:

    * Prior surgery for an aneurysm;
    * Have cardiac pacemaker;
    * Have metal fragments in the eyes, brain, or spinal cord from shrapnel, metal work, or welding;
    * Have surgical implants, such as ear implant or neurostimulator;
    * Have a history of claustrophobia;
    * Have a history of not tolerating previous MRI scans without medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J Irrgang, PT, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were referred to the study by their athletic trainer and/or physician at the UPMC Center for Sports Medicine/ University of Pittsburgh between July 2016 and December 2022. The first participant was enrolled on August 10, 2016, and the last participant was enrolled on August 4, 2021.
Pre-assignment Details: Of the 183 individuals with hamstring injuries screened for the study, 17 met the inclusion/exclusion criteria and were eligible for the study. Nine of the eligible individuals declined to consent, and 8 agreed to consent. Two participants withdrew from the study prior to randomization, leaving 6 participants randomized to treatment.
Groups:
- Losartan: Subjects took 50mg of Losartan per day for 4 weeks.
- Placebo: Subjects were given a placebo to replicate the appearance of Losartan pills. Placebo pill was taken once per day.
Period: Overall Study
Arm/Group | Losartan | Placebo
Started | 3 | 3
Week 1 Follow-up | 3 | 3
Week 2 Follow-up | 3 | 3
Week 3 Follow-up | 3 | 3
Week 4 Follow-up | 3 | 3
Week 6 Follow-up | 2 | 3
3 Month Follow-up | 2 | 3
6 Month Follow-up | 2 | 3
9 Month Follow-up | 2 | 3
12 Month Follow-up | 2 | 2
Completed | 2 | 2
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 32 [21 to 47] | 21.7 [21 to 22] | 26.8 [21 to 47]
Age, Customized [Count of Participants; unit: Participants]
  Age: 21 years old | 1 | 1 | 2
  Age: 22 years old | 0 | 2 | 2
  Age: 28 years old | 1 | 0 | 1
  Age: 47 years old | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.5 (3.0) | 28.6 (4.2) | 28.5 (3.3)
Side of Injury [Count of Participants; unit: Participants]
  Left | 2 | 2 | 4
  Right | 1 | 1 | 2
Primary Sport [Count of Participants; unit: Participants] — Sport individual was playing at time of injury
  Participants
    Baseball | 0 | 1 | 1
    Football | 1 | 2 | 3
    Soccer | 1 | 0 | 1
    Tennis | 1 | 0 | 1
Extent of the initial injury: Proximal-distal length [Mean (Full Range); unit: centimeters] — Magnetic Resonance Imaging (MRI) evaluation of the proximal-distal length of the initial injury
  centimeters | 23.0 [12.7 to 32.6] | 21.8 [18.4 to 28.0] | 22.4 [12.7 to 32.6]
Extent of the initial injury: Volume of injury [Mean (Full Range); unit: cubic centimeters] — Magnetic Resonance Imaging (MRI) evaluation of the volume of initial injury
  cubic centimeters | 588.4 [50.2 to 1576.0] | 816.8 [267.5 to 1789] | 702.6 [50.2 to 1789]

OUTCOME MEASURES:

1. Primary Outcome: Reported Effects of Losartan for Hamstring Injury for Safety and Tolerability
Description: Directly related to specific aim 1- Side effects, safety, and tolerability will be monitored by measuring vital signs, lab values via blood work, and number of adverse events, serious adverse events, and patient reported side effects.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 3 | 3
Participants
  Hypotension | 0 | 0
  Serious adverse events | 0 | 0
  Drug related adverse event | 0 | 0
  Side effects | 0 | 0
  Abnormal labs | 0 | 0
  No adverse events, serious adverse events, and patient reported side effects. | 3 | 3

2. Primary Outcome: Recovery of Hamstring Muscle Function
Description: For specific aim 2, hamstring muscle function of the injured leg was measured and compared to the contralateral leg using isometric hamstring force at 30, 60, and 90 degrees of knee flexion at 6 weeks and 6 months.
  Data are expressed as a Limb Symmetry Index (LSI), which is the percent force of the injured hamstring compared to the force of the non-injured hamstring muscle.
Time Frame: 6 weeks; 6 months
Population: Losartan Group: 4 wk data at 30 & 90 degrees substituted for 6 wk data (1 subject lost to follow-up at 4 wks, 1 data not collected). 6 wk data at 60 degrees missing for subject lost to follow-up at 4 wks. 6 m data missing for subject lost to follow-up at 4 wks & not collected for 1 subject Placebo group: 6 wk data at 60 degrees not collected for 1 participant. 6 m data missing for 1 subject that moved out of the area prior to 6 m & data not collected for 1 subject at 60 degrees of flexion
Measure: Mean (95% Confidence Interval); unit: % of contralateral limb strength
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 3 | 3
% of contralateral limb strength
  6 weeks: Limb Symmetry Index isometric strength at 30 deg knee flexion (Handheld dynamometer) | 91 [42 to 139] | 75 [21 to 129]
  6 weeks: Limb Symmetry Index isometric strength at 90 deg knee flexion (Handheld dynamometer) | 102 [67 to 137] | 77 [69 to 85]
  6 weeks: Limb Symmetry Index isometric strength at 60 deg knee flexion (Biodex): number analyzed (Participants) | 2 | 2
  6 weeks: Limb Symmetry Index isometric strength at 60 deg knee flexion (Biodex) | 79 [59 to 98] | 73 [15 to 130]
  6 months: Limb Symmetry Index isometric strength at 30 deg knee flexion (Handheld dynamometer): number analyzed (Participants) | 2 | 2
  6 months: Limb Symmetry Index isometric strength at 30 deg knee flexion (Handheld dynamometer) | 107 [0 to 323] | 95 [0 to 355]
  6 months: Limb Symmetry Index isometric strength at 90 deg knee flexion (Handheld dynamometer): number analyzed (Participants) | 2 | 2
  6 months: Limb Symmetry Index isometric strength at 90 deg knee flexion (Handheld dynamometer) | 106 [0 to 290] | 76 [0 to 590]
  6 months: Limb Symmetry Index isometric strength at 60 deg knee flexion (%, Biodex): number analyzed (Participants) | 2 | 1
  6 months: Limb Symmetry Index isometric strength at 60 deg knee flexion (%, Biodex) | 83 [45 to 121] | 104

3. Primary Outcome: Recovery of Hamstring Structure
Description: For specific aim 2, recovery of hamstring structure was measured as the length of injury at 6 months as well as the change in proximal-distal length of injury from baseline to 6 month post-treatment MRI. Greater change in length represents greater healing.
Time Frame: 6 months
Population: Losartan group: one participant was completely lost to follow-up after 4 weeks. There is also missing MRI data for 6-month timepoint for one other participant.
  Placebo group: one participant moved out of the area before the 6-month visit and did not complete the 6 month clinical research visit.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 1 | 2
centimeters
  Proximal-distal length of injury measured (MRI) | 0.8 | 5.6 [0 to 67]
  Change in proximal-distal length of injury from baseline (MRI) | 23 | 17.6 [0 to 140]

4. Primary Outcome: Recovery of Hamstring Structure
Description: For specific aim 2, hamstring structure was measured in terms of the volume of fibrosis at 6 month MRI, as such smaller volume of fibrosis represents greater healing of the hamstring muscle. Hamstring structure was also determined by comparing the change of pre-treatment volume of the injury on the baseline MRI to the volume of fibrosis on the 6 month MRI.
Time Frame: 6 months
Population: Losartan group: one participant was completely lost to follow-up after 4 weeks. There is also missing MRI data for 6-month timepoint for one other participant.
  Placebo group: one participant moved out of the area before the 6-month visit and did not complete the clinical research visit.
Measure: Mean (95% Confidence Interval); unit: cubic centimeters
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 1 | 2
cubic centimeters
  Volume of fibrosis at 6 months (MRI) | 0.6 | 0.7 [0 to 3]
  Change of pre-treatment volume of the injury to 6 months (MRI) | 138.4 | 1028 [0 to 10691]

5. Primary Outcome: Return to Prior Level of Function
Description: Return to prior level of function will be measured by the number of days from injury to full, unrestricted return to practice. This could have occurred at any timepoint after 6 weeks, so this did not necessarily occur at 12 months but it was monitored until the 12 month timepoint.
Time Frame: 12 months
Population: Despite losing one participant in the Losartan group after 4 weeks and one in the placebo group after 9 months, data for this outcome was able to be collected and analyzed as the participants returned to their prior level of function before they were lost to follow-up.
Measure: Mean (Full Range); unit: days
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 3 | 3
days | 23 [14 to 42] | 35 [7 to 70]

6. Primary Outcome: Recurrence of Injury
Description: Number of recurrent injuries will be monitored during the duration of the subjects participation.
Time Frame: 12 months
Population: Losartan group: one participant was completely lost to follow-up after 4 weeks. Placebo group: one participant moved out of the area before the 6-month visit and did not complete the clinical assessment portion, however reinjury reporting was tracked until 9 months, after which the individual was lost to further follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 2 | 3
Participants
  Recurrent hamstring injury | 0 | 2
  No recurrent hamstring injury | 2 | 1

7. Secondary Outcome: Recovery of Hamstring Structure
Description: For specific aim 2, restoration of hamstring structure was operationally defined as the ratio of the volume of the injured to contralateral leg hamstring volume 6 months after injury 6 months post-injury. The percent of hamstring volume of the injured leg was expressed as a percentage of the hamstring volume of the contralateral normal leg. The difference in volume between the involved and non-involved hamstring muscles was divided by the non-involved hamstring muscle volume and multiplied by 100.
Time Frame: 6 months
Population: Losartan group: one participant was completely lost to follow-up after 4 weeks. There is also missing MRI data for 6-month timepoint for one other participant.
  Placebo group: one participant moved out of the area before the 6-month visit and did not complete the clinical research follow-up visit and then was completely lost to follow-up after the 9 month telephone call.
Measure: Mean (95% Confidence Interval); unit: Percent of contralateral hamstring vol
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 1 | 2
Percent of contralateral hamstring vol | 0.91 | 3.9 [-2.8 to 10.7]

8. Secondary Outcome: Return to Prior Level of Function
Description: For specific aims 3 and 4, return to prior level of sports activity was measured by the Marx Activity Scale Score, which ranges from 0 to 16, with 16 being the highest level of sports activity. The frequency of participants who achieved the same or better Marx score at follow-up compared to baseline was calculated. Differences from baseline to each follow-up timepoint were calculated by subtracting the follow-up scores from baseline. Any difference of 0 or a negative number indicated the participants achieved the same level of sports activity or better. Positive differences indicated they did not return to their prior level of sports activity.
Time Frame: 4 Weeks, 6 Weeks, 3 Months, 4 Months, 6 Months, 12 Months
Population: Losartan group: one participant was completely lost to follow-up after 4 weeks. Placebo group: one participant moved out of the area before the 6-month visit and did not complete the clinical assessment portion of the research follow-up, then was completely lost to follow-up after the 9 month telephone call.
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 3 | 3
Participants
  Marx Activity Level Score: Achieved prior level or better at 4 Weeks | 1 | 1
  Marx Activity Level Score: Achieved prior level or better at 6 Weeks: number analyzed (Participants) | 2 | 3
  Marx Activity Level Score: Achieved prior level or better at 6 Weeks | 1 | 1
  Marx Activity Level Score: Achieved prior level or better at 3 Months: number analyzed (Participants) | 2 | 3
  Marx Activity Level Score: Achieved prior level or better at 3 Months | 2 | 3
  Marx Activity Level Score: Achieved prior level or better at 4 Months: number analyzed (Participants) | 2 | 3
  Marx Activity Level Score: Achieved prior level or better at 4 Months | 1 | 3
  Marx Activity Level Score: Achieved prior level or better at 6 Months: number analyzed (Participants) | 2 | 2
  Marx Activity Level Score: Achieved prior level or better at 6 Months | 1 | 1
  Marx Activity Level Score: Achieved prior level or better at 12 Months: number analyzed (Participants) | 2 | 2
  Marx Activity Level Score: Achieved prior level or better at 12 Months | 1 | 1

9. Secondary Outcome: Recovery of Hamstring Flexibility
Description: For specific aim 2, hamstring muscle flexibility of the injured leg was measured and compared to the contralateral leg using the popliteal angle at 6 weeks and 6 months after randomization. The popliteal angle was measured with a goniometer. Recovery of hamstring flexibility was operationally defined as the difference in the popliteal angle between the contralateral normal leg minus the hamstring injured leg. Positive differences between the contralateral and injured leg indicated decreased hamstring flexibility.
Time Frame: 6 weeks; 6 months
Population: Losartan group: one participant was completely lost to follow-up after 4 weeks. Placebo group: one participant moved out of the area before the 6-month visit and did not complete the clinical research follow-up and then was completely lost to follow-up after the 9 month telephone call.
Measure: Mean (95% Confidence Interval); unit: difference in degrees of popliteal angle
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 2 | 3
difference in degrees of popliteal angle
  Difference in popliteal angle between injured and non-injured limb at 6 weeks | 1.0 [-11.7 to 13.7] | -1.3 [-7.1 to 4.4]
  Difference in popliteal angle between injured and non-injured limb at 6 months: number analyzed (Participants) | 2 | 2
  Difference in popliteal angle between injured and non-injured limb at 6 months | -1.5 [-20.6 to 17.6] | -0.5 [-6.9 to 5.9]

10. Secondary Outcome: Recovery of Hamstring Muscle Function
Description: For specific aim 2, hamstring muscle function of the injured leg was measured and compared to the contralateral leg using isometric hamstring force at 1 week, 2 weeks, 3 weeks, and 4 weeks. Data were expressed as a Limb Symmetry Index (LSI), which is the percent strength of the injured hamstring in comparison to the strength of the non-injured hamstring muscle.
Time Frame: 1 week; 2 weeks; 3 week; 4 weeks
Population: For the 4 week strength assessment, one participant in the Losartan group did not have isometric strength testing completed.
Measure: Mean (95% Confidence Interval); unit: % of contralateral limb strength
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 3 | 3
% of contralateral limb strength
  1 week: Limb Symmetry Index isometric strength at 30 deg knee flexion (Handheld dynamometer) | 70.8 [0.3 to 141.2] | 54.9 [-37.2 to 147.1]
  1 week: Limb Symmetry Index isometric strength at 90 deg knee flexion (Handheld dynamometer) | 83.9 [62.2 to 105.6] | 39.8 [-59.7 to 139.2]
  2 weeks: Limb Symmetry Index isometric strength at 30 deg knee flexion (Handheld dynamometer) | 83.3 [39.8 to 126.8] | 50.1 [28.8 to 71.4]
  2 weeks: Limb Symmetry Index isometric strength at 90 deg knee flexion (Handheld dynamometer) | 93.8 [60.1 to 127.5] | 44.6 [23.1 to 66.2]
  3 weeks: Limb Symmetry Index isometric strength at 30 deg knee flexion (Handheld dynamometer) | 103.0 [-24.1 to 230.2] | 87.2 [47.9 to 126.4]
  3 weeks: Limb Symmetry Index isometric strength at 90 deg knee flexion (Handheld dynamometer) | 95.9 [-0.7 to 192.5] | 69.1 [-1.3 to 139.4]
  4 weeks: Limb Symmetry Index isometric strength at 30 deg knee flexion (Handheld dynamometer): number analyzed (Participants) | 2 | 3
  4 weeks: Limb Symmetry Index isometric strength at 30 deg knee flexion (Handheld dynamometer) | 79.1 [45.6 to 112.7] | 82.5 [44.2 to 120.7]
  4 weeks: Limb Symmetry Index isometric strength at 90 deg knee flexion (Handheld dynamometer): number analyzed (Participants) | 2 | 3
  4 weeks: Limb Symmetry Index isometric strength at 90 deg knee flexion (Handheld dynamometer) | 106.5 [-35.3 to 248.3] | 91.6 [69.0 to 114.1]

11. Secondary Outcome: Recovery of Hamstring Muscle Function
Description: For specific aim 2, hamstring muscle function of the injured leg was measured on the Biodex and compared to the contralateral leg using isokinetic peak torque at 60 degrees and 180 degrees per second at 6 weeks and 6 months. Data were expressed as a Limb Symmetry Index (LSI), which is the percent peak torque of the injured hamstring compared to the peak torque of the non-injured hamstring muscle.
  The isokinetic testing was not consistently collected, so there are limited results to present at 6 months.
Time Frame: 6 weeks, 6 months
Population: Losartan group: At 6 weeks, one participant was completely lost to follow-up after 4 weeks, and another participant did not complete isokinetic testing. At 6 months, data was collected for one participant, since one was lost to follow-up and the other did not complete isokinetic testing.
  Placebo group: At 6 weeks, data is missing for one participant, and another did not complete isokinetic testing. At 6 months, data was not collected for this group.
Measure: Mean (95% Confidence Interval); unit: % of contralateral limb peak torque
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 1 | 1
% of contralateral limb peak torque
  6 Weeks: Limb Symmetry Index isokinetic peak torque at 60 deg per second (Biodex) | 96.5 | 202.7
  6 Weeks: Limb Symmetry Index isokinetic peak torque at 180 deg per second (Biodex) | 104.1 | 71.2
  6 Months: Limb Symmetry Index isokinetic peak torque at 60 deg per second (Biodex): number analyzed (Participants) | 1 | 0
  6 Months: Limb Symmetry Index isokinetic peak torque at 60 deg per second (Biodex) | 105.3 |
  6 Months: Limb Symmetry Index isokinetic peak torque at 180 deg per second (Biodex): number analyzed (Participants) | 1 | 0
  6 Months: Limb Symmetry Index isokinetic peak torque at 180 deg per second (Biodex) | 81.3 |

12. Secondary Outcome: Recovery of Hamstring Muscle Function
Description: For specific aim 2, hamstring muscle function of the injured leg was measured on the Biodex and compared to the contralateral leg using isokinetic total hamstring work at 60 degrees per second and 180 degrees per second at 6 weeks and 6 months. Data were expressed as a Limb Symmetry Index (LSI), which is the percent total work of the injured hamstring compared to the total work of the non-injured hamstring muscle.
  The isokinetic testing was not consistently collected, so there are limited results to present at 6 months.
Time Frame: 6 weeks, 6 months
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: % of contralateral limb total work
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 1 | 1
% of contralateral limb total work
  6 Weeks: Limb Symmetry Index isokinetic total hamstring work at 60 deg per second (Biodex) | 108.9 | 484.2
  6 Weeks: Limb Symmetry Index isokinetic total hamstring work at 180 deg per second (Biodex) | 134.2 | 63.3
  6 Months: Limb Symmetry Index isokinetic total hamstring work at 60 deg per second (Biodex): number analyzed (Participants) | 1 | 0
  6 Months: Limb Symmetry Index isokinetic total hamstring work at 60 deg per second (Biodex) | 113.8 |
  6 Months: Limb Symmetry Index isokinetic total hamstring work at 180 deg per second (Biodex): number analyzed (Participants) | 1 | 0
  6 Months: Limb Symmetry Index isokinetic total hamstring work at 180 deg per second (Biodex) | 78.9 |

13. Secondary Outcome: Recovery of Hamstring Muscle Function
Description: For specific aim 2, the ratio of hamstring peak torque to quadriceps peak torque at 60 degrees per second of the injured and non-injured legs were measured on the Biodex at 6 weeks.
  The isokinetic testing was not consistently collected, so there are limited results to present at 6 months.
Time Frame: 6 weeks, 6 months
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: ratio of hams. to quad. peak torque
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 1 | 1
ratio of hams. to quad. peak torque
  6 Weeks: Ratio of hamstring peak torque to quadriceps peak torque at 60 deg per second | 51.9 | 33.9
  6 Months: Ratio of hamstring peak torque to quadriceps peak torque at 60 deg per second: number analyzed (Participants) | 1 | 0
  6 Months: Ratio of hamstring peak torque to quadriceps peak torque at 60 deg per second | 70.7 |

14. Secondary Outcome: Recovery of Hamstring Muscle Function
Description: For specific aim 2, the ratio of hamstring work in the last 3 repetitions to work in the first 3 repetitions at 180 degrees per second of the injured leg was measured on the Biodex at 6 weeks.
  The isokinetic testing was not consistently collected, so there are no results to present at 6 months.
Time Frame: 6 weeks, 6 months
Population: Losartan group: At 6 weeks, one participant was completely lost to follow-up after 4 weeks, and another participant did not complete isokinetic testing.
  Placebo group: At 6 weeks, data is missing for one participant, and another did not complete isokinetic testing.
  Data was not collected at 6 months for either group.
Measure: Mean (95% Confidence Interval); unit: ratio of work in last 3 to first 3 reps
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 1 | 1
ratio of work in last 3 to first 3 reps | 153.1 | 76.7

ADVERSE EVENTS:
Time Frame: 12 months
Description: During the 4 week period of active intervention while taking the Losartan or placebo, subjects were followed weekly with activity level and adverse event monitoring and blood pressure measurements. Activity level and adverse event monitoring also occurred via telephone follow-up at 12 weeks and 4, 9, and 12 months. Blood pressure was also evaluated at 6 weeks and 6 months. Blood work (and pregnancy tests for women) was assessed at 2, 4, and 6 weeks after randomization.
Arm/Group | Losartan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=3) | Placebo (N=3)
Hamstring reinjury (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Recruitment was complicated primarily due to delays in identifying potential study participants, as individuals were often excluded for presenting > 7 days from injury (n=106), not having at least a grade 2 injury (n=9), or refusing participation (n=9). The study was terminated due to the expiration of funding, which resulted in a sample size of 6 participants. Given this sample size was smaller than anticipated, no between-group significance testing was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-03-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT02263729/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT02263729/ICF_001.pdf